CLINICAL TRIAL: NCT02268682
Title: Improving Low-Income End Stage Renal Disease Patients' Transplant Knowledge: A Case Management Trial
Brief Title: Explore Transplant at Home: Improving Low-Income ESRD Patients' Transplant Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Missouri Kidney Program (Unknown)
Responsible Party: Principal Investigator, Amy D. Waterman, Director, Patient Engagement, Diversity, and Education, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R39OT26843
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: End Stage Renal Disease
Keywords: Educator-Guided; Patient-Guided; Standard of Care (Control)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of Care (Control) (No Intervention): Patients randomized to the standard of care condition will not receive any educational materials from our program and will only participate in the survey portion of the investigation. Dialysis providers will be asked to continue their current practices throughout the study period without change. While Control patients will be free to ask additional questions or solicit more information from their dialysis educators at any point during the study period, no additional educational interventions will be added to what is currently being done.
- Patient-Guided (Experimental): Over an 8-month period, patients in the Patient-Guided intervention condition will receive four educational modules and twelve transplant education postcards in the mail. Modules will be mailed once every other month and consist of an introductory letter, a transplant video, and printed resources. Transplant education postcard will be mailed every two weeks following the mailing of each module, for a total of three postcards over the course of 6-weeks.
  Interventions: Other: Patient-Guided
- Educator-Guided (Experimental): Patients in the Educator-Guided intervention condition will receive the same intervention components as those in the Patient-Guided condition; however, the key difference in this condition is that Educator-Guided patients will also receive telephonic support from an experienced clinical social worker in the role of a Transplant Educator to maximally facilitate learning. Telephonic meetings with the Transplant Educator will occur after the mailing of each study module, for a total of four calls, each lasting 20-minutes, totaling 1 hour and 20 minutes. Finally, Patient-Guided and Educator-Guided patients will have the option of enrolling in an educational text messaging service designed to supplement the ET education they are receiving in the mail.
  Interventions: Other: Patient-Guided; Other: Educator-Guided

INTERVENTIONS:
Other: Patient-Guided — The "Explore Transplant" education program was designed to increase patient informed decision-making and knowledge and is based on the theoretical tenets of the Transtheoretical Model of Behavior Change. The program helps patients think about what might motivate them to pursue transplant, addresses commonly held concerns about transplant and involving a living donor, and shares real-life transplant stories of donors and recipients. The ET materials were written for patients with low health literacy. Already developed for the "Explore Transplant" program are brochures, videos, and factsheets. ET at Home is an expansion of the ET program. Newly designed postcards and text messages have added to the list of transplant education resources for this program.
  Other Names: Explore Transplant at Home
  Arms: Educator-Guided; Patient-Guided
Other: Educator-Guided — The Transplant Educator supports the Explore Transplant at Home materials by facilitating a conversation about the content of the materials. The role of the Educator is filled by an experienced dialysis healthcare provider who can support a patient as they learn about their treatment options. The program is split into a series of four modules and the Educator conversations are guided by a Transplant Educator Guide and Patient Tracking Tool. This tool is intended to provide direct talking points for the Educator and is also a place where the patients' responses, questions, or concerns can be documented.
  Other Names: Transplant Educator
  Arms: Educator-Guided

SUMMARY:
Kidney transplantation, especially living donor kidney transplant (LDKT), offers patients in end-stage renal disease (ESRD) 3 to 17 additional years of life and improved quality-of-life compared to remaining on dialysis. Unfortunately, LDKT education in dialysis centers occurs inconsistently, especially for minorities and those who are socioeconomically disadvantaged.

To ensure more informed transplant decision-making, through a previous HRSA grant, Dr. Waterman designed the Explore Transplant (ET) education program based on the Transtheoretical Model of Behavioral Change. Through a previous trial, an earlier version of ET, delivered face-to-face with patients while they were undergoing dialysis, was shown to increase patients' DDKT and LDKT knowledge. However, additional research exploring dialysis providers' ability to integrate ET into their care revealed that multiple patient, provider, and system barriers limited the degree to which transplant education could be improved.

Thus, a more comprehensive case-management program to educate patients through external organizations may be needed to supplement ongoing transplant education within dialysis centers. For this grant, the investigators propose to test the effectiveness of another replicable solution for disseminating ET education on a broad scale: Partnering with a large health insurance organization to deliver video-guided transplant education supported by telephone and mail. The Missouri Kidney Program (MoKP) is a state-wide organization whose mission is to serve and educate kidney patients, particularly those who are economically disadvantaged. Since MoKP subsidizes the costs of dialysis medication for low-income ESRD patients, they operate as an insurance company would with respect to their 1200-patient member group. With 900 dialysis patients currently being managed by the MoKP, the investigators will conduct an eight-month, group randomized controlled trial (GRCT) where 540 patients will be randomized to receive: (1) no additional education other than from their dialysis center; (2) a video-guided, four-part Explore Transplant (ET) program delivered via the internet or mail; or (3) a video-guided ET program with discussion facilitated by a telephone case manager.

DETAILED DESCRIPTION:
Nationwide, there are almost 600,000 patients with end-stage renal disease (ESRD), or kidney failure. There are two options for ESRD patients to sustain life: dialysis, where a machine filters wastes from the blood, or a kidney transplant from a deceased or living donor. Kidney transplantation, especially living donor kidney transplant (LDKT), offers ESRD patients 3 to 17 additional years of life and improved quality-of-life compared to remaining on dialysis.

However, the majority of ESRD patients- 415,000 as of 2009 - still remain on dialysis. Although dialysis is life-saving, it only replaces 10-15% of normal kidney function and can lead to cardiovascular disease, infection, and other complications. Dialysis treatment also takes 12 to 15 hours per week, requiring many patients to stop work and go on disability. The chance of a dialysis patient being alive after 5 years without a transplant is only 38%.

A complex set of potential risks and benefits need to be considered when deciding whether to get an LDKT, particularly for low-income dialysis patients facing significant practical and financial barriers to transplant. Established chronic kidney disease (CKD) and Centers for Medicaid and Medicare Services (CMS) guidelines recommend that dialysis patients be educated about their different treatment options, the medical risks involved, and the advantages to transplant so that they can make informed transplant decisions. Since transplants within the first six months of beginning dialysis result in the best health outcomes, one Healthy People 2020 proposed goal is to, "Increase the proportion of dialysis patients wait-listed and/or receiving a deceased donor kidney transplant within one year of ESRD start (among patients under 70 years of age)". Unfortunately, research has shown that many patients in dialysis centers are inconsistently educated about LDKT, particularly patients who are socioeconomically disadvantaged or members of racial/ethnic minority groups.

Through a previous HRSA grant, Dr. Waterman designed the Explore Transplant (ET) education program based on Prochaska's Transtheoretical Model of Behavioral Change and her own research with over 1000 patients with kidney disease to address key gaps in patients' transplant knowledge. The mission of ET is for transplant-eligible patients to explore the option of transplant and make an informed choice after knowing the benefits and risks. Through a group randomized controlled trial (GRCT), an earlier version of ET, delivered face-to-face with patients while they were undergoing dialysis, was shown to increase patients' knowledge and informed decision-making. As a result, the Explore Transplant program won the 2009 National Association of Transplant Professionals (NATCO) Quality of Care Award. However, additional research exploring dialysis providers' ability to integrate ET in their patient care found that multiple patient, provider, and system barriers limited what can be accomplished educationally within dialysis centers. With dialysis providers reporting that they have limited time to educate patients, a more comprehensive case-management program through external organizations may be needed to supplement the inconsistent transplant education provided within dialysis centers.

Thus, for this grant, the investigators propose to test the effectiveness of another replicable and transferable solution for disseminating ET transplant education nationally for patients in chronic kidney disease (CKD) Stages 3-5: Partnering with a large health insurance organization to provide transplant education supported by telephone and mail. The important research question now requiring study is whether this dissemination strategy also can promote greater transplant knowledge for patients, particularly for the most vulnerable patients least likely to receive comprehensive transplant education from dialysis centers.

For this grant, the investigators have chosen to re-partner with an organization with which the investigators have had previous success conducting transplant education trials, the Missouri Kidney Program (MoKP). Since MoKP subsidizes the costs of dialysis and transplant medication for low-income ESRD patients in Missouri, they operate as an insurance company would with respect to their 1200-patient member group. MoKP is also a natural ally for underserved groups of kidney patients and can focus on educating them comprehensively about DDKT and LDKT without other competing job responsibilities. Finally, they have strong, statewide partnerships with every dialysis center in Missouri, with permission to communicate with social workers about the needs, transplant education needs and care of specific dialysis patients.

Therefore, in partnership with the MoKP, this grant team will conduct a group randomized controlled trial (GRCT) of 540 low-income dialysis patients in order to assess how an established, video-guided transplant education program, Explore Transplant, could be incorporated within a centralized health care organization's delivery of transplant education. The investigators will conduct an eight-month educational intervention where patients will be randomized to receive: (1) no additional education other than what is provided within the dialysis center; (2) a video-guided, four-part ET program delivered via the internet or mail; or (3) a video-guided, four-part ET program with discussion facilitated by a Transplant Educator via telephone. The investigators expect 20% attrition over time for a final sample of 430 Black and White patients. The investigators will also conduct considerable formative work to assess the unique difficulties faced by Black and White low-income patients in learning about transplant online and by telephone.

The grant aims are:

Aim 1: To understand the transplant educational needs and barriers to learning faced by low-income Black and White ESRD patients.

Aim 2: Compared to standard-of-care dialysis center education, to conduct a GRCT to assess the effectiveness of patient-guided and case-manager-guided ET education on improving low-income patients' DDKT and LDKT knowledge and informed LDKT decision-making.

Aim 3: To examine how patient characteristics and the quality of their dialysis center transplant education act alone and in combination with the ET educational programs

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following inclusion criteria to be enrolled:

1. Participant must be 18-74 years of age.
2. Participant must self-identify as African American or White.
3. Participant must currently be on dialysis.
4. Participant must have a household income at or below 250% of the federal poverty level.
5. Participant must be able to speak and read in English.

Exclusion Criteria:

Subjects that meet any of the following exclusion criteria are not to be enrolled:

1. Participant has a visual and/or hearing impairment that would preclude him/her from watching and reading educational study material.
2. Participant has had a previous kidney transplant
3. Participant has previously been told that they are not a candidate for transplant.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Deceased Donor Kidney Transplant (DDKT) and Living Donor Kidney Transplant (DDKT) Knowledge | 9 months
  Patients will be asked 17 true/false and 8 multiple choice questions to determine their level of knowledge regarding basic facts, advantages, risks and outcomes of DDKT and LDKT (e.g., "Patients older than 75 years can receive transplants"; "Compared to transplants from donors who have died, how long do transplants from living donors last?"). Scores for this scale are created by summing the number of correct answers given by the patient, creating a theoretical range of 0-25 with higher scores indicating more knowledge.

SECONDARY OUTCOMES:
Informed Decision-Making | 9 months
  Informed Decision-Making will be assessed in two ways. First, patients will be asked the following three questions: "I have all the facts I need to make an informed decision about whether to pursue DDKT/LKDT/remain on dialysis" (agree/disagree). Each of these questions will be treated as individual items and analyzed separately as outcomes.
  We will also use a validated measure of decisional conflict, the Decisional Conflict Scale (DCS). This scale assesses factors contributing to patients' uncertainty in making health-related decisions, and patients' assessment of their perceived effective decision-making. Each of these dimensions of decisional conflict will be considered as subscales, and together they will be considered as a total decisional conflict measure. The entire scale has 16 items (3 for decision uncertainty, 9 for factors contributing to uncertainty, and 4 for effective decision-making), each measured on a scale of (1) strongly agree to (5) strongly disagree. Total scale
Decisional Balance | 9 months
  Decisional Balance will be measured for DDKT (DB-DDKT) and for LDKT (DB-LDKT). DB-DDKT, a measure of a patient's perception of the benefits and disadvantages of deceased donor kidney transplant. This measure has been validated in a sample of dialysis patients84. Both measures contain two subscales, Pros and Cons of 6 items, wherein patients rate the importance of a specific Pro or Con to their DDKT or LDKT decision-making (e.g., "I would not have to be on dialysis") on a Likert-type scale from (1) "Not important" to (5) "Extremely important". Scores for the subscales will be obtained by summing the patients' responses to the items, implying a theoretical range of 6-30, with higher scores indicating more Pros or Cons, depending on the subscale. The DB-LDKT was also recently validated in a sample of dialysis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Waterman, PHD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Transplant Research and Education Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waterman AD, Peipert JD, McSorley AM, Goalby CJ, Beaumont JL, Peace L. Direct Delivery of Kidney Transplant Education to Black and Low-Income Patients Receiving Dialysis: A Randomized Controlled Trial. Am J Kidney Dis. 2019 Nov;74(5):640-649. doi: 10.1053/j.ajkd.2019.03.430. Epub 2019 Jun 19. PMID 31227225
- [Derived] Waterman AD, McSorley AM, Peipert JD, Goalby CJ, Peace LJ, Lutz PA, Thein JL. Explore Transplant at Home: a randomized control trial of an educational intervention to increase transplant knowledge for Black and White socioeconomically disadvantaged dialysis patients. BMC Nephrol. 2015 Aug 28;16:150. doi: 10.1186/s12882-015-0143-0. PMID 26316264